CLINICAL TRIAL: NCT00698854
Title: A Prospective, Non-controlled, Clinical Investigation of the Vanguard™ Complete Knee System
Brief Title: A Clinical Investigation of the Vanguard™ Complete Knee System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.K005
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis; Traumatic Arthritis; Rheumatoid Arthritis; Lower Limb Deformity; Complications, Arthroplasty
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vanguard™ Complete Knee System: Vanguard Total Knee System, Cruciate-Retaining (CR) or Posterior-Stabilized (PS)
  Interventions: Device: Vanguard™ Complete Knee System
- Vanguard™ Patient-Specific Femur: Vanguard Total Knee System used in combination with Signature technique to provide a patient-specific femur
  Interventions: Device: Vanguard™ Patient-Specific Femur

INTERVENTIONS:
Device: Vanguard™ Complete Knee System — Primary Total Knee System, Cruciate-Retaining (CR) or Posterior-Stabilized (PS)
  Groups: Vanguard™ Complete Knee System
Device: Vanguard™ Patient-Specific Femur — Primary Total Knee System used with Signature technique to provide a patient-specific femur
  Other Names: Vanguard Select
  Groups: Vanguard™ Patient-Specific Femur

SUMMARY:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of the Vanguard™ Complete Knee System.

DETAILED DESCRIPTION:
This is a 10-year prospective observational data collection on the Vanguard Total Knee system. Patients are asked to come in for a preop, operative, immediate post-operative, 6 Month, 1 Year, 3 Year,5 Year, 7 year, and 10 year visits to check on the function, range of motion, and radiographic assessment of their total knee device.

The Vanguard Knee is an FDA cleared device, and has been on the market since 2004.

ELIGIBILITY:
Inclusion criteria:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity
* Correction or revision of unsuccessful osteotomy, or arthrodesis

Patient selection factors to be considered include:

* Need to obtain pain relief and improve function
* Ability and willingness of the patient to follow instructions
* Including control of weight and activity level
* Good nutritional state of the patient
* Patient must have reached full skeletal maturity

Exclusion criteria:

Absolute contraindications include:

* Infection
* Sepsis
* Osteomyelitis
* Failure of a previous joint replacement

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, Muscular atrophy, Neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee

Additional exclusion criteria includes: failure of a previous joint replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of relief from painful or disabling joint disease
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2004-03; Primary Completion 2021-01 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
KSS | 10 year
  Knee Society Score Assessment

SECONDARY OUTCOMES:
Radiographic Information | 10 years
  Radiographic Evaluation Report
Survivorship | 10 years
  Knee Society Score Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Kacy C Arnold, RN MBA, Study Director — Zimmer Biomet
Locations (8):
- United States (8):
  - Physicians Clinic of Iowa Orthopedics, Cedar Rapids, Iowa
  - The Orthopaedic Center, Rockville, Maryland
  - Advanced Orthopedic Specialists, Cape Girardeau, Missouri
  - Orthopaedic Associates of Rochester, Rochester, New York
  - Texas Orthopedic Specialists, Grapevine, Texas
  - Orthopedic Associates, Fishersville, Virginia
  - Spokane Orthopedics, Spokane, Washington
  - Othopaedic & Sports Medicine Clinic of Monroe, Monroe, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided